CLINICAL TRIAL: NCT04391465
Title: Assessment of the Relationship Between Cerebral Blood Flow and Heart Rate: An Electrophysiology Based Study
Brief Title: Assessment of the Relationship Between Cerebral Blood Flow and Heart Rate
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REB20-0064
Record Dates: First submitted 2020-03-22; First posted 2020-05-18 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Cerebrovascular Circulation; Physiology
Keywords: Cerebral Blood Flow

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients Scheduled for Elective Electrophysiological Study (Experimental): High right atrial pacing will occur at the following rates for 60 seconds each, with a rest period of at least 60 seconds between pacing runs:
  * 600 msec (100 bpm)
  * 500 msec (120 bpm)
  * 400 msec (150 bpm)
  * 350 msec (171 bpm)
  Interventions: Other: Electrophysiological Pacing

INTERVENTIONS:
Other: Electrophysiological Pacing — Assess the MCA CBF velocity response at different paced heart rates.

SUMMARY:
The investigators will seek to determine the relationship between heart rate and middle cerebral artery (MCA) cerebral blood flow (CBF), as well as better understand the hemodynamic determinants of MCA CBF velocity. In order to manipulate heart rate, the investigators will recruit patients already scheduled for clinically indicated elective electrophysiological studies, where temporary pacing catheters placed in the right atrium can be used to artificially pace the heart at controlled rates. MCA CBF will be measured by transcranial Doppler ultrasound.

DETAILED DESCRIPTION:
Background: Cerebral blood flow (CBF) is maintained at a relatively constant level by multiple overlapping auto-regulatory systems over a wide range of blood pressures. This ensures adequate oxygen delivery to the brain and is critical to ongoing brain function and consciousness. Patients with reduced CBF experience symptoms of presyncope (e.g. lightheadedness, dizziness, trouble concentrating) and may faint. In patients with postural tachycardia syndrome (POTS), these orthostatic symptoms are a chronic issue, but the underlying pathophysiology is poorly understood - there is both evidence for and against impaired cerebral auto-regulation in POTS patients.

Previous studies have demonstrated that increased cardiac output improves CBF independent of mean blood pressure. This is of particular interest in POTS patients, who display reduced cardiac output both during rest and orthostasis. This is due in part smaller heart size and reduced blood volume, which necessitate high heart rates to maintain cardiac output. The relationship between cardiac output and CBF has not been studied in POTS patients. Given the characteristic orthostatic tachycardia seen in these patients, the effects of heart rate on CBF are also of interest. The relationship between heart rate and CBF, to our knowledge, has not been studied.

The chronic orthostatic symptoms in POTS patients are largely unexplained, but contributed centrally to significantly reduced quality of life. These symptoms are thought to be caused in part by alterations in CBF. While POTS does not have a "cure", alleviation of orthostatic symptoms would likely improve patients' ability to engage with activities of daily living and may reduce overall disease burden. Gaining an improved understanding of the hemodynamic determinants of CBF is essential to achieving this goal.

Objectives: To assess the relationship between heart rate and middle cerebral artery (MCA) CBF. Additionally, to better understand the hemodynamic determinants of MCA CBF velocity by examining the relationships between heart rate, stroke volume, pulse pressure, and MCA CBF velocity.

Methods: This will be an open-label, single group study in otherwise healthy patients scheduled for elective electrophysiology studies prior to planned ablations for supraventricular tachycardia. The study will take place with the participant supine on the electrophysiology laboratory procedure table, with a temporary pacing catheter already placed in the high right atrium. Prior to beginning the study protocol, the participant will be instrumented with non-invasive (a) skin electrodes to continuously monitor heart rate and record an electrocardiogram; (b) a volume-clamp finger cuff to monitor beat-to-beat blood pressure, calibrated with intermittent brachial cuff measurements; and (c) a transcranial Doppler System to record CBF velocity. Estimates of stroke volume, cardiac output, and systemic vascular resistance will be obtained using Modelflow-based waveform analysis of the continuous blood pressure waveform. A clinically standard sinus node recovery time (SNRT) protocol will be performed whilst collecting CBF and hemodynamic responses. Pacing will occur at 600 ms (100 bpm), 500 ms (120 bpm), 400 ms (150 bpm), and 350 ms (171 bpm) cycles for 60 seconds each, with a rest period of at least 60 seconds between pacing runs. After these pacing runs, the study data collection will be complete and the extra blood pressure cuffs and transcranial doppler probes will be removed from the participant so that the clinical electrophysiology study may continue as planned. The investigators estimate that this study will add no more than 10-15 minutes to the overall procedure time.

In this exploratory "proof of concept" study, the investigators plan to enrol 20 participants.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Age 18-70 years, inclusive
* Scheduled for clinically indicated elective electrophysiological studies where temporary pacing catheters are being placed in the right atrium
* Left ventricular ejection fraction ≥50%
* Able and willing to provide informed consent
* Able to travel to the Cardiac Electrophysiology Laboratory at the Foothills Medical Centre, Calgary, Alberta, Canada

Exclusion Criteria:

* Unable or unwilling to provide informed consent
* Other factors which in the investigator's opinion would prevent the participant from completing the protocol

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-08-11 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Change in MCA CBF velocity in response to high right atrial pacing at 400 ms (150 bpm) relative to baseline while in the supine position | After 1 minute of pacing at 400 ms (150 bpm)
  Compare the MCA CBF velocity at the participant's own baseline sinus rhythm (<100 bpm) and during pacing at 400 ms (150 bpm)

SECONDARY OUTCOMES:
Change in MCA CBF velocity in response to high right atrial pacing at 600 ms (100 bpm) relative to baseline while in the supine position | After 1 minute of pacing at 600 ms (100 bpm)
  Compare the MCA CBF velocity at the participant's own baseline sinus rhythm (<100 bpm) and during pacing at 600 ms (100 bpm)
Change in MCA CBF velocity in response to high right atrial pacing at 350 ms (171 bpm) relative to baseline while in the supine position | After 1 minute of pacing at 350 ms (171 bpm)
  Compare the MCA CBF velocity at the participant's own baseline sinus rhythm (<100 bpm) and during pacing at 350 ms (171 bpm)
Change in MCA CBF velocity in response to high right atrial pacing at 400 ms (150 bpm) relative to pacing at the lowest rate (100 bpm) while in the supine position | 10 minute electrophysiological pacing protocol
  Compare the MCA CBF velocity during pacing at 600 ms (100 bpm) and during pacing at 400 ms (150 bpm)
Change in MCA CBF velocity in response to high right atrial pacing at 350 ms (171 bpm) relative to pacing at the lowest rate (100 bpm) while in the supine position | 10 minute electrophysiological pacing protocol
  Compare the MCA CBF velocity during pacing at 600 ms (100 bpm) and during pacing at 350 ms (171 bpm)
Change in stroke volume in response to high right atrial pacing at 400 ms (150 bpm) relative to baseline while in the supine position | 10 minute electrophysiological pacing protocol
  Compare the stroke volume at the participant's own baseline sinus rhythm (<100 bpm) and during pacing at 400 ms (150 bpm)
Change in cardiac output in response to high right atrial pacing at 400 ms (150 bpm) relative to baseline while in the supine position | 10 minute electrophysiological pacing protocol
  Compare the cardiac output at the participant's own baseline sinus rhythm (<100 bpm) and during pacing at 400 ms (150 bpm)
Change in pulse pressure in response to high right atrial pacing at 400 ms (150 bpm) relative to baseline while in the supine position | 10 minute electrophysiological pacing protocol
  Compare the pulse pressure at the participant's own baseline sinus rhythm (<100 bpm) and during pacing at 400 ms (150 bpm)

CONTACTS AND LOCATIONS:
Overall Officials: Satish R Raj, MD MSCI, Principal Investigator — University of Calgary
Locations (1):
- Foothills Medical Center, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No